CLINICAL TRIAL: NCT06735066
Title: Effects of Abnormalities of Preoperative Ascending Urethrocystography on the Short-term Outcomes of Living Donor Kidney Transplantation
Brief Title: Abnormalities of Preoperative Ascending Urethrocystography and Outcomes of Living Donor Kidney Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shehabeldin Alaa Ahmed Mahmoud Ahmed Saad, resident doctor at Urology department Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: Kidney transplantation 2024
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplantation
Keywords: preoperative ascending urethrocystography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Transplantation group: adult patients who underwent kidney transplantation
  Interventions: Procedure: Ascending urethrocystography

INTERVENTIONS:
Procedure: Ascending urethrocystography — It will be performed after instructing the patient to evacuate the bladder. A contrast agent will be infused through the urethra under fluoroscopy, using a urethral catheter or Knutson's clamp at the external urethral meatus. When the bladder is full, an anteroposterior film and two oblique films will be taken. Voiding cystourethrography will be performed as a part of this imaging examination. From this procedure, the following findings may be diagnosed:
  * Upper urinary tract: Vesicoureteral reflux (VUR); laterality and degrees of VUR will be defined.
  * Bladder: Capacity (defunctionalized, Small-sized or contracted bladder), neurogenic bladder, bladder diverticulum, filling defects, etc.
  * Urethra: Stricture and filling defects.

SUMMARY:
To evaluate effects of abnormalities in preoperative ascending urethrocystography on the short-term outcomes of LDKT

DETAILED DESCRIPTION:
The incidence of surgical complications after kidney transplantation (KT) has decreased in recent decades due to improvements in surgical techniques and immunosuppression protocols. However, the preoperative abnormalities of the urinary tract may influence the outcomes of KT. Hence, the preoperative evaluation of the urinary tract is a critical step in the KT process to identify the potential risk factors for poor outcomes .

Ascending urethrocystography (AUC) is a key diagnostic tool to assess the integrity and functionality of the lower urinary tract . It provides detailed insights into the bladder, urethra, vesicoureteral valves, and surrounding structures, identifying any abnormalities that could pose risks during or after KT . Understanding this issue is crucial, as certain urological anomalies may predispose patients to complications such as urinary leaks, infections, or delayed graft function, potentially leading to poorer short-term outcomes .

Although AUC is used indiscriminately as a screening test for urological abnormalities, only 6% of all KT recipients may have abnormal lower urinary tract . Few studies have looked at the yield from AUC and attempted to assess objectively whether certain patients could be selected for KT based on a positive result in AUC . Accordingly, the impact of abnormalities detected in AUC on the short-term outcomes of living donor KT (LDKT) remains inefficiently studied .

This is the rationale to conduct this cohort study on patients undergoing LDKT. We hypothesize that the presence of abnormalities in AUC will influence the surgical outcomes and short-term survival rates after LDKT

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult patients undergoing LDKT in Assiut Kidney Transplantation Unit.
* Patients with preoperative evaluation by AUC.

Exclusion Criteria:

* Patients with a primary non-functioning graft after LDKT.
* Patients with missing relevant preoperative or postoperative data.
* Patients refusal to participate in the study.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult patients who underwent kidney transplantation
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of urinary complications post kidney transplantation | 6 month
  Each patient will be followed up for the surgical complications for 6- month duration after KT

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] John EE, Mehta S, Sohal PM, Sandhu JS. Predictors of Short-Term Outcomes in Living Donor Renal Allograft Recipients: A Prospective Study From a Tertiary Care Center in North India. Cureus. 2022 Aug 24;14(8):e28335. doi: 10.7759/cureus.28335. eCollection 2022 Aug. PMID 36168334
- [Background] Jayanth ST, Dangi AD, Mukha RP, Kumar S, Varughese S, David VG, Valson A, Chandrasingh J, Devasia A, Kekre N. Renal transplantation into optimized abnormal lower urinary tract - Impact on graft outcomes, patient survival, and complications. Indian J Urol. 2019 Jan-Mar;35(1):67-72. doi: 10.4103/iju.IJU_203_18. PMID 30692727
- [Background] Freitas PS, Alves AS, Correia PS, Dias JL. Urethrocystography: a guide for urological surgery? Diagn Interv Radiol. 2023 Jan 31;29(1):9-17. doi: 10.5152/dir.2022.21640. Epub 2022 Dec 21. PMID 36959709
- [Background] Sellers MT, Velidedeoglu E, Bloom RD, Grossman RA, Markmann JW, Naji A, Frank AM, Kass AB, Nathan HM, Hasz RD, Abrams JD, Markmann JF. Expanded-criteria donor kidneys: a single-center clinical and short-term financial analysis--cause for concern in retransplantation. Transplantation. 2004 Dec 15;78(11):1670-5. doi: 10.1097/01.tp.0000144330.84573.66. PMID 15591958